CLINICAL TRIAL: NCT01618435
Title: The Clinical Effect of i-FACTOR® Versus Allograft in Non-instrumented Posterolateral Spondylodesis Operation
Brief Title: The Clinical Effect of i-FACTOR® Versus Allograft in Non-instrumented Posterolateral Spondylodesis Operation in the Elderly With Spinal Stenosis Due to Degenerative Spondylolisthesis
Acronym: IVANOS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sygehus Lillebaelt (Other)
Collaborators: CeraPedics, Inc (Industry)
Responsible Party: Principal Investigator, Michael Kjaer Jacobsen, MD, Sygehus Lillebaelt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F12-04
Record Dates: First submitted 2012-05-08; First posted 2012-06-13 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Spinal Stenosis
Keywords: Fusion surgery; Degenerative olisthesis; i-FACTOR; ODI; Spinal stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Fibrinogen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fusion, allograft (Active Comparator): Allograft used for fusion in the operation site
  Interventions: Biological: i-FACTOR
- Fusion, i-FACTOR (Experimental): i-FACTOR used for fusion in the operation site
  Interventions: Biological: i-FACTOR

INTERVENTIONS:
Biological: i-FACTOR — i-FACTOR mixed with autologous bone from the decompression placed in the operation site for enhancing fusion
  Other Names: i-FACTOR®putty, Cerapedics, USA. CE-brand 0086

SUMMARY:
The average life expectancy in Denmark is increasing resulting in an increasing part of the population having age-related disease, ex lumbar spinal stenosis (LSS). LSS causes constriction of the nerves in the lumbar spine resulting in pain in the legs and lower back, especially when standing and walking, known as neurogenic claudication(Goh KJ FAU - Khalifa et al.). LSS occurs in a combination of degenerative changes in the lower back, including hypertrophy of the ligamentum flavus, arthrosis of the facet joints and bulging of the disc.

Current treatment of LSS is varied ranging from non-operative conservative treatment to operation.

Operative intervention shows very good results according to physical ability and pain(Christensen FB et al.;Hee HT and Wong;McGregor AH FAU - Hughes and Hughes;Xu et al.), but the most optimal treatment is still debated. Nevertheless, a decompression and, if needed, a spinal fusion is recommended.(Ausman).

Clinical improvement including decrease of pain, improved ADL-function and an increased quality of life are parameters of highest interest and the purpose of an operation is clear: Making sufficient room for the affected nerves. In addition fusion is desired achieving stability avoiding a new compression of the nerves. Studies attending these issues find a correlation between fusion and clinical outcome, why obtained fusion of the affected levels are very important(Andersen et al.;Andersen et al.;Girardo et al.;Kornblum MB FAU - Fischgrund et al.).

P-15, bound to Anorganisk Bone Mineral (ABM), called i-FACTOR®, shows fusion superiority, no side effects and no risk of transferring disease(Thorwarth et al. 5648-57;Thorwarth et al. 789-95;Wenz, Oesch, and Horst 1599-606;Scarano et al. 318-24;Kubler et al. 171-79) why the investigators find this material suited for fusion surgery in the elderly.

To the investigators knowledge this is the first prospective study comparing fusion rates and postoperative clinic with i-FACTOR vs allograft in older patients operated with decompression and spondylodesis because of spinal stenosis due to degenerative spondylolisthesis.

Hypothesis:

There are no difference in the clinical parameters measured by ODI and fusion rates comparing i-FACTOR® and allograft in non-instrumented posterolateral spondylodesis-operations in patients 60 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Spinal stenosis, olisthesis grade 1-2 (>3 mm), facet joint arthrosis and flavus hypertrophia verified by a mr-scan and x-ray including maximally 2 levels ranging from L1-S1.
* A score of 6 and more on Konno´s "History of Examination Characteristic".
* Signed informed content.

Exclusion Criteria:

* Any disease demanding obligate thromboprophylaxis treatment, including mechanical valve, (DVT with cancer/thrombophilia, AMI, apoplexia cerebri, TCI, valve-operation)< 3 months, coronar metal stent < 6 weeks and coronar drug eluted/coated stent < 12 months.
* Atrial fibrillation and one of the following: Mitral stenosis, valveprothesis and apoplexia cerebri/TCI.
* Atrial fibrillation and two of the following: Heart insufficient, HT, DM, age > 75 years, EF < 35 %.
* Known cancer in the axial skeleton.
* Ongoing chemotherapy.
* Fracture i the lower back within a year prior to inclusion.
* Reduced distance of walking due to non-spinal related causes.
* Candidate for more than two-level intervention.
* Dementia assessed by the MMSE
* ASA 3+4
* Age below 60 years.
* Missed 3 months of conservative treatment without success
* The use of steroids and bisphosphonates.
* Prior radiotherapy to the lower back.
* Haematologic disease.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
The clinical effect of i-FACTOR® versus allograft in non-instrumented posterolateral spondylodesis operation in the elderly with spinal stenosis due to degenerative spondylolisthesis measured by ODI | 24 months postoperative

SECONDARY OUTCOMES:
The clinical effect of i-FACTOR® versus allograft in non-instrumented posterolateral spondylodesis operation in the elderly with spinal stenosis due to degenerative spondylolisthesis assessed by fusion rates | 12 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Michael K Jacobsen, MD, Principal Investigator — Rygkirurgisk sektor Middelfart
Locations (2):
- Denmark (2):
  - Sygehuslillebaelt, Middelfart, DK
  - Rygkirurgisk sektor Middelfart, Middelfart, Region Syddanmark